CLINICAL TRIAL: NCT02584348
Title: Ultrasound Assessment of Gastric Contents : the Way to Best Induce Children for Emergency Surgery
Brief Title: Gastric Ultrasound in Paediatric Anaesthesia
Acronym: ECHOGASTRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013.790
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: General Anesthesia
Keywords: ultrasound, antrum, pulmonary aspiration, emergency surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gastric Ultrasound (Experimental): Preoperative qualitative ultrasound assessment of gastric contents will be performed
  Interventions: Device: Gastric ultrasound

INTERVENTIONS:
Device: Gastric ultrasound — Preoperative qualitative ultrasound assessment of gastric contents will be performed for each children admitted for emergency surgery

SUMMARY:
Anesthesia for emergency surgery is a situation at risk of pulmonary aspiration of gastric contents. It has been previously reported that bedside two-dimensional ultrasonography can be a useful tool for anesthesiologists to determine gastric contents and volume in adults and children.

In this prospective study, preoperative qualitative ultrasound assessment of gastric contents is performed for each children admitted for emergency surgery, in order to plane in case of empty stomach an intravenous or inhalation technique induction rather than an rapid sequence induction.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 0 to 18 years old
* Parental consent

Exclusion Criteria:

* Gastric tube contraindication
* Parental refusal

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 146 (Actual)
Dates: Start 2013-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of adapted changes in induction technique according to ultrasound assessment of gastric contents | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Dominique CHASSARD, MD, PhD, Principal Investigator — Department of paediatric anaesthesia, Hôpital Femme Mère Enfant, Hospices Civils de Lyon
Locations (1):
- Department of paediatric anaesthesia, Bron, France

REFERENCES:
- [Result] Gagey AC, de Queiroz Siqueira M, Monard C, Combet S, Cogniat B, Desgranges FP, Robinson P, Chassard D, Bouvet L. The effect of pre-operative gastric ultrasound examination on the choice of general anaesthetic induction technique for non-elective paediatric surgery. A prospective cohort study. Anaesthesia. 2018 Mar;73(3):304-312. doi: 10.1111/anae.14179. Epub 2017 Dec 19. PMID 29265174